

## Royal Brompton & Harefield **NHS**



## **PARTICIPANT CONSENT FORM**

| NAWI | E OF PARTICIPANT: | ••••• | *************************************** | |
|---|---|---|---|---|
| | of the project: A cross-section ssment in surgical coronary reva | - | el screening survey for ra | adial artery |
| Main i | investigator and contact details: | Vincenzo De Franco | vincenzo.de-franco@po | gr.aru.ac.uk |
| 1. | I agree to take part in the all Information Sheet (Date 23 Mathematical What my role will be in this answered to my satisfaction. | May 2024 V 5.0) for | the study. I understand | Please initia |
| 2. | I understand that I am free to withdraw from the research at any time, without giving a reason, by speaking with the researcher or emailing them at <a href="mailto:vincenzo.de-franco@pgr.aru.ac.uk">vincenzo.de-franco@pgr.aru.ac.uk</a> stating the title of the research. Data collected up until the point of withdrawal may still be used in analysis. | | | |
| 3. | I am free to ask any questions at any time before and during the study. | | | |
| 4. | I understand what information will be collected from me for the study. | | | |
| 5. | For the purposes of the Data Protection Act (2018), if this project requires me to produce personal data, I have read and understood how Anglia Ruskin University and will process it. | | | |
| 6. | I understand that some information will be collected from existing records held about me. | | | |
| 7. | I understand what will happen to the data collected from me for the research. | | | |
| 8. | I have been informed how my data will be processed, how long it will be kept and when it will be destroyed. | | | |
| 9. | I understand that I will be provided with summary of the findings. | | | |
| 10. | I have been provided with a copy of this form and the Participant Information Sheet (Date 23 May 2024 V 5.0). | | | |
| | Name of participant | Date | Signature | |
| Name of researcher | | Date | Signature | |

PARTICIPANTS MUST BE GIVEN A COPY OF THIS FORM TO KEEP

Date 23 May 2024 Version 5.0